CLINICAL TRIAL: NCT03075358
Title: Effects of Lidocaine Spray for Reducing Pain During Endometrial Aspiration Biopsy : a Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OBG-2559-04137
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Uterine Bleeding
MeSH Terms: conditions — Uterine Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine spray (Experimental)
  Interventions: Drug: Lidocaine spray
- Normal saline spray (Sham Comparator)
  Interventions: Other: Normal saline spray
- No spray (No Intervention)

INTERVENTIONS:
Drug: Lidocaine spray — Patients are locally anesthetized with 8 puffs (80 mg, 10mg/puff, 0.8 ml) of 10% lidocaine spray applied thoroughly to the cervix, 3 minutes before starting the procedure.
  Arms: Lidocaine spray
Other: Normal saline spray — 0.8 ml of normal saline spray is applied to the cervix, 3 minutes before starting the procedure
  Arms: Normal saline spray

SUMMARY:
Endometrial aspiration biopsy has been accepted as a diagnostic procedure of choice for women with abnormal uterine bleeding to examine endometrial pathology. The procedure has high accuracy comparing to conventional fractional curettage. However, it is associated with significant pain during the procedure. In general, there is no specific recommendation regarding the proper anesthesia used during the procedure.

The aim of this study is to examine the effect of lidocaine spray for reducing pain during the endometrial aspiration procedure by comparing it with placebo and no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing endometrial aspiration biopsy at Maharaj Nakorn Chiang Mai hospital

Exclusion Criteria:

* Lidocaine allergy
* Pregnancy
* Previous uterine or cervical surgical procedures
* Neurological abnormalities
* Coagulopathy
* Infection of cervix, vagina, or pelvic cavity
* Taking any analgesic drugs within 4 hours before the procedure

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Aspiration pain | Immediately following endometrial aspiration biopsy
  A visual analog scale pain score associated with endometrial aspiration biopsy
Postprocedure pain | 10 minute after procedure completion
  A visual analog scale pain score after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Study Chair — Faculty of Medicine, Chiang Mai University; Ratpaporn Piyawetchakarn, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided